CLINICAL TRIAL: NCT06938347
Title: A Phase 3, Open-label, Multicenter, Randomized Crossover Trial Comparing the Safety and Efficacy of ASI-02 to Agitated Saline for Suspected Right-to-left Shunt
Brief Title: Comparing the Safety and Efficacy of ASI-02 to Agitated Saline for Suspected Right-to-left Shunt
Acronym: ENHANCE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Agitated Solutions, Inc. (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ASI-CL-0301
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Right-To-Left Shunt
Keywords: Saline Contrast; Saline Contrast Transthoracic Echocardiogram; Transthoracic Echocardiogram; Agitated Saline Standard of Care; Echocardiogram; Transpulmonary Shunt

STUDY DESIGN:
Intervention Model Description: For each participant, the first two (2) injections will be agitated saline SoC (one [1] injection at rest, one [1] injection during a maneuver). Next, participants will be randomized to either receive two (2) ASI-02 injections followed by two (2) agitated saline SoC injections, or vice versa (with each pair involving an injection at rest and an injection during a maneuver).
Who Masked: Outcomes Assessor
Masking Description: This is an open-label study; therefore, blinding procedures are not necessary for site personnel or participants. Blinded assessment of the primary efficacy endpoint will be completed by the core lab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care to ASI-02 TTE Study (Experimental): Participants will be allocated to a saline contrast echocardiography study with agitated saline SoC, followed by a saline contrast echocardiography study with ASI-02.
  Interventions: Drug: Agitated Saline SoC; Drug: ASI-02
- ASI-02 to Standard of Care TTE Study (Experimental): Participants will be allocated to a saline contrast echocardiography study with ASI-02, followed by a saline contrast echocardiography study with agitated saline SoC.
  Interventions: Drug: Agitated Saline SoC; Drug: ASI-02

INTERVENTIONS:
Drug: Agitated Saline SoC — The recommended initial dose of agitated saline SoC is approximately 10 mL of saline containing approximately 1 mL of air, per institutional policy, rapidly mixed (approximately 10-20 presses) to manufacture microbubbles. No additives are allowed to the saline, including blood, dextrose, or bacteriostatic saline.
Drug: ASI-02 — Each injection shall utilize one (1) ASI-02 product connected to one (1) pre-filled 10 mL 0.9% sodium chloride (saline) syringe. The ASI-02 investigational product will be connected to a standard luer lock connector and administered in its entirety. The intravenous bolus injected dose of ASI-02 is 9 mL of saline and 1 mL of air.

SUMMARY:
This is a phase 3, multicenter, open-label, blinded, crossover trial in which each participant will undergo a randomized sequence of ASI-02 and agitated saline standard of care (SoC) via a saline contrast transthoracic echocardiogram (TTE) study.

DETAILED DESCRIPTION:
The primary objective is to determine the safety of ASI-02 and its agreement with agitated saline SoC for detection of right-to-left shunt in saline contrast studies utilizing TTE in the intended setting of use (opacifying the right heart). The investigation will be conducted in up to 8 investigational sites in the U.S. and Canada. Participants will receive n=2 ASI-02, n=4 agitated saline SoC injections as part of a single-day imaging session, with the overall duration for study participation of 24 to 48 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is clinically indicated for a saline contrast TTE study with a suspected right-to-left shunt
2. Patient must be at least 18 years of age inclusive, at the time of signing the informed consent
3. Able to communicate effectively with trial personnel

Exclusion Criteria:

1. Female patients who are pregnant or lactating. All women of child-bearing potential (WOCBP) must have a negative urine pregnancy test at screening regardless of contraceptive use history
2. WOCBP are excluded unless they have been using an adequate and medically approved method of contraception to avoid pregnancy for at least 1 month prior to ASI-02 dose administration
3. Allergy to polysorbate 80 (PS-80)
4. American Society of Anesthesiologists (ASA) physical status classification IV, V, or VI, except that participants with ASA physical status IV due solely to recent suspected transient ischemic attack or cerebrovascular accident are eligible for inclusion
5. Current illness or pathology that in the opinion of the investigator would prevent undergoing investigational product administration due to a significant safety risk to the patient
6. Uncontrolled arterial hypertension (defined as systolic blood pressure ≥ 200 mmHg or diastolic blood pressure ≥ 110 mmHg) or arterial hypotension (defined as systolic blood pressure ≤ 90 mmHg)
7. Unstable cardiovascular status defined as:

   1. myocardial infarction or unstable angina pectoris within 6 months prior to procedure day
   2. symptomatic valvular heart disease or moderate to severe stenotic valvular heart disease
   3. clinically significant congenital heart defects (excluding an atrial septal defect [ASD], patent foramen ovale [PFO], or pulmonary arteriovenous malformation [PAVM])
   4. current uncontrolled cardiac arrhythmias causing clinical symptoms requiring medical intervention or hemodynamic compromise
   5. acute pulmonary embolus or pulmonary infarction
   6. acute myocarditis or pericarditis
   7. acute aortic dissection
   8. untreated atrial fibrillation
8. Any major surgery within 30 days prior to screening
9. Participation in any investigational drug, device, or placebo study within 30 days prior to screening
10. Vulnerable adult participant populations (e.g., incarcerated or cognitively challenged adults)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Positive percentage agreement (PPA) of ASI-02 for detecting right-to-left shunt versus agitated saline SoC | Procedure through 24- to 48-hour participant follow-up visit
Negative percentage agreement (NPA) of ASI-02 for detecting right-to-left shunt versus agitated saline SoC | Procedure through 24- to 48-hour participant follow-up visit

SECONDARY OUTCOMES:
The incidence of ASI-02-related adverse events | 24- to 48-hour participant follow-up visit
Peak opacification intensity | Procedure through 24- to 48-hour participant follow-up visit
Contrast opacification duration | Procedure through 24- to 48-hour participant follow-up visit
Positive percentage agreement (PPA) of ASI-02 for shunt detection at rest | Procedure through 24- to 48-hour participant follow-up visit
Negative percentage agreement (NPA) of ASI-02 for shunt detection at rest | Procedure through 24- to 48-hour participant follow-up visit
Positive percentage agreement (PPA) of ASI-02 for shunt detection specific to shunt sizes | Procedure through 24- to 48-hour participant follow-up visit
Negative percentage agreement (NPA) of ASI-02 for shunt detection specific to shunt sizes | Procedure through 24- to 48-hour participant follow-up visit
Test-retest reliability of agitated saline SoC | Procedure through 24- to 48-hour participant follow-up visit
Positive percentage agreement (PPA) of ASI-02 for detecting right-to-left shunt versus agitated saline SoC, using the first (nonrandomized) SoC study. | Procedure through 24- to 48-hour participant follow-up visit
Negative percentage agreement (NPA) of ASI-02 for detecting right-to-left shunt versus agitated saline SoC, using the first (nonrandomized) SoC study. | Procedure through 24- to 48-hour participant follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Narang, MD, Principal Investigator — Northwestern Medicine
Locations (5):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - NYU Langone Health, New York, New York
- Toronto General, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No
Due to the potential risks to participant privacy, the possibility of re-identification, concerns about data misuse for commercial purposes, and the potential harm to participants due to sensitive health information, IPD will not be available to other researchers.